CLINICAL TRIAL: NCT06302361
Title: Lymphovenous Anastomosis for Breast Cancer-related Lymphedema: A Cohort Study
Brief Title: Lymphovenous Anastomosis for Breast Cancer Lymphedema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Vejle Hospital (Other); Zealand University Hospital (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Caroline Lilja, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/54225
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Lymphedema; Lymphedema Arm; Breast Cancer Lymphedema; Lymphedema, Secondary; Lymphedema; Surgical; Lymphedema of Upper Limb; Lymphedema, Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Cancer Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Multi-center cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphovenous anastomosis (LVA) (Experimental): Intervention with lymphovenous anastomosis (LVA) surgery of the affected arm.
  Interventions: Procedure: Lymphovenous anastomosis (LVA)

INTERVENTIONS:
Procedure: Lymphovenous anastomosis (LVA) — Surgical procedure with supermicrosurgical anastomosis between distal lymph vessel and proximal venule.
  Other Names: Lymphovenous bypass; Lymphaticovenular anastomosis

SUMMARY:
This multi-center cohort study focuses on evaluating the efficacy of lymphovenous anastomosis (LVA) for treating pitting lymphedema in female breast cancer survivors. Conducted across multiple centers in Denmark, including Odense University Hospital, Herlev Hospital, Lillebaelt Hospital Vejle, and Zealand University Hospital, it aims to assess LVA's impact on reducing arm volume and improving quality of life in patients with upper extremity lymphedema secondary to breast cancer treatment.

Eligible participants are adult women with unilateral arm lymphedema who show active pitting and identifiable lymphatic vessels via indocyanine green lymphography. Inclusion involves informed consent and the ability to complete Danish questionnaires.

Patients are recruited from the outpatient clinics of the participating hospitals and will undergo LVA surgery under either local or general anesthesia. Following the intervention, patients are seen for data collection up to twelve months.

The study measures outcomes like arm volume changes through water displacement volumetry and arm circumferential measurements, body composition via bioimpedance, health-related quality of life through LYMPH-Q, general quality of life through SF-36, arm function via DASH, and anastomosis patency via ICG lymphography. Additionally, changes in ICG lymphography images, arm fibrosis via SkinFibroMeter, and surgery duration are evaluated.

The study adheres to ethical guidelines, ensuring patient safety and the integrity of the research.

DETAILED DESCRIPTION:
This comprehensive single-armed cohort study is dedicated to assessing the effectiveness of lymphovenous anastomosis (LVA) in treating pitting lymphedema among adult female patients who have undergone breast cancer treatment.

This study builds upon findings from our preliminary pilot study at Odense University Hospital, and is conducted across several hospitalt in Denmark, including Odense University Hospital, Lillebælt Hospital Vejle, Zealand University Hospital Roskilde, and Herlev Hospital.

The study's primary aim is to determine whether LVA can significantly reduce arm volume and improve the overall quality of life for patients afflicted with breast cancer-related lymphedema.

Inclusion Criteria and Patient Recruitment The study population consists of women over 18 years of age suffering from unilateral arm lymphedema secondary to breast cancer treatment. Key eligibility criteria include active pitting lymphedema, presence of dermal backflow as evidenced by indocyanine green lymphography, identifiable lymphatic vessels in the affected arm, and the ability to provide informed consent and complete questionnaires in Danish.

Prospective participants are identified during clinical assessments at the participating hospitals' Departments of Plastic Surgery. Those deemed suitable for LVA surgery by consulting surgeons are invited to participate, ensuring informed consent through both oral and written communication.

Method This multi-center cohort study employs a range of outcome measures to evaluate the impact of LVA surgery. Primary outcomes focus on changes in arm volume, measured through water displacement volumetry and arm circumferential measurements, employing the unaffected arm as a control.

Secondary outcomes include assessments of body composition via bioimpedance spectroscopy, health-related quality of life through the LYMPH-Q questionnaire, arm function via the DASH questionnaire, general quality of life via the SF-36 questionnaire, patency of anastomosis validated by ICG lymphography, changes in ICG lymphography images, and arm fibrosis measured with the SkinFibroMeter.

Data collected are entered into a secure database for analysis. This includes comparing pre- and postoperative measurements to assess the primary and secondary outcomes.

Surgical Procedure and Follow-up LVA surgeries are performed by surgeons at Odense University Hospital and Herlev Hospital, with the choice between local or general anesthesia based on the number of planned anastomoses and patient preference.

Patients will be seen prior to surgery for baseline measurements, in addition to six and twelve months post-operative follow-up. At three and nine months post-operative, phone consultations will be performed for reminders of questionnaires and patient safety.

The study prohibits participants from undergoing other medical or surgical treatments for lymphedema during the trial period, although conservative treatments like compression garments are accepted.

Data Management and Ethics Adhering to the ethical standards, this study complies with Good Clinical Practice, The Danish Code of Conduct for Research Integrity, and GDPR. It has sought approval from the Research Ethics Committee of the Region of Southern Denmark. Patient safety is paramount, with LVA considered a safe and valid treatment option.

Feasibility and Publication Led by Caroline Lilja, MD, and Ph.D. student, under the supervision of Jørn Bo Thomsen, Dr., MD., Ass. Prof., the study aims for results publication regardless of the outcome, emphasizing its contribution to the field and potential impact on treatment protocols for lymphedema patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Female
* Unilateral arm lymphedema secondary to breast-cancer treatment
* Active pitting lymphedema
* Presence of dermal backflow in indocyanine green lymphography
* Identifiable lymphatic vessel(s) in the affected arm using an infrared camera and indocyanin green
* Able to provide informed consent
* Able to read, understand and complete Danish questionnaires

Exclusion Criteria:

* Allergy to iodine
* Pregnant, breast-feeding, or aiming to conceive withing the next year
* History of bilateral breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Arm volume (Water Displacement) | Baseline, six months, twelve months
  Changes of arm volume difference
Arm volume (Arm Circumferences) | Baseline, six months, twelve months
  Changes of arm volume difference

SECONDARY OUTCOMES:
Health-related quality of life (LYMPH-Q) | baseline, three months, six months, nine months, twelve months
  Changes of health-related quality of life, measured with LYMPH-Q
General quality of life (SF-36) | baseline, three months, six months, nine months, twelve months
  Changes of health-related quality of life measured with SF-36
Arm and shoulder function (DASH) | baseline, three months, six months, nine months, twelve months
  Changes in arm and shoulder function, measured with DASH
L-Dex | Baseline, six months, twelve months
  Changes in L-Dex score
LVA patency | Baseline, six months
  Evaluation of patency using indocyanine green lymphography postoperatively. Number of patent anastomosis will be compared to number performed during surgery.
Skin Fibrosis | Baseline, six months, twelve months
  The degree of skin fibrosis measured with SkinFibroMeter
Surgery duration | Day of intervention
  The duration of surgery will be compared between sites
Body composition | Baseline, six months, twelve months
  Changes in body compositions measured with SoZo bioimpedance will be evaluated.
Skin Water Content | Baseline, six months, twelve months
  The water content in the dermis measured with LymphScanner

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Lilja, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Plastic Surgery, Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT06302361/Prot_SAP_000.pdf